CLINICAL TRIAL: NCT03642184
Title: Efficacy and Safety of Empagliflozin Compared With Linagliptin in New-onset Diabetes Mellitus After Kidney Transplantation
Brief Title: Efficacy and Safety of Empagliflozin in NODAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult in enrolling suitable participants
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ20180601NODAT
Record Dates: First submitted 2018-07-16; First posted 2018-08-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: New Onset Diabetes After Transplant; Kidney Transplant; Complications
Keywords: empagliflozin; linagliptin; diabetes; kidney transplantation
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin; Linagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin (Active Comparator): Jardiance 10mg/25mg Film-coated tablets， once daily
  Interventions: Drug: Empagliflozin
- Linagliptin (Active Comparator): Trajenta 5mg Film-coated tablets， once daily
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Empagliflozin — Dosage adjustment based on glucose targets . Once daily
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Linagliptin — Dosage adjustment based on glucose targets. Once daily
  Other Names: Tradjenta
  Arms: Linagliptin

SUMMARY:
This is an open label, randomized controlled study. We'd like to access the safety and effects of empagliflozin compared with linagliptin in new-onset diabetes after kidney transplantation patients. Our primary endpoints are kidney related indicators and secondary endpoints are glucose and lipid metabolism related indicators and adverse events. We are going to recruit 35 patients for each group and follow six months.

DETAILED DESCRIPTION:
In recent years, with the development of transplantation technology and immunosuppressive agents, kidney transplantation has made considerable progress. However, for metabolic disorders after kidney transplantation, such as new diabetes after kidney transplantation, there is still insufficient awareness. Since 1964, Starlz et al. first discovered and proposed New-onset diabetes after kidney transplantation（NODAT） in patients after renal transplantation. Scholars from all countries have paid considerable attention to it. The Chinese guidelines indicate that NODAT can increase the risk of graft-related complications, such as rejection, graft loss and infection, and ultimately affect the long-term survival of the recipient. In addition, NODAT has also been shown to increase the risk of cardiovascular events, and cardiovascular disease is associated with more than half of kidney transplant deaths. A retrospective study of 567 renal transplant recipients in China showed that the incidence of NODAT was 24.2%. It can be seen that the incidence of new-onset diabetes after renal transplantation is high and has long-term adverse effects on transplant patients. Therefore, there is an urgent need to evaluate and investigate NODAT's therapeutic drug regimens.

According to the study, empagliflozin has a protective effect on the kidney and cardiovascular system, but it has not yet been written into the treatment guidelines for new-onset diabetes after kidney transplantation. Metformin and linagliptin are frequently used in diabetics after renal transplantation, and linagliptin also have a protective effect on the kidneys. Therefore, this experiment wanted to compare the effects between empagliflozin and linagliptin on kidney protection.

ELIGIBILITY:
Inclusion Criteria:

* Single kidney transplantation
* Normal glucose tolerance or Pre-Diabetes mellitus before transplantation
* According to Oral glucose tolerance test results to make the diagnosis of NODAT
* Standard triple immunosuppression therapy
* HbA1c≤10%
* Steady hormone usage
* BMI 18.5-30kg/m2
* Patient informed consent

Exclusion Criteria:

* Diabetes patients before transplantation
* Pregnancy pregnancy
* Type 1 diabetes after kidney transplantation
* Severe liver function impairment (AST/ALT 3 times standard value)
* Severely impaired renal function (eGFR<45)
* Having uncontrolled diseases
* History of cancer in the past 5 years (except basal cell carcinoma) and/or cancer treatment
* Participating in another trial involving the study drug with in 30 days
* Premenopausal women (1 year before the last menstrual period ≤ informed consent)
* Alcohol or drug abuse within 3 months of informed consent, affecting compliance Need other drugs to control NODAT

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
eGFR | 24 weeks
  the change from baseline in estimated glomerular filtration rate calculated by MDRD formula

SECONDARY OUTCOMES:
Graft loss rate | 24 weeks
  the frequency of patients' graft loss or dysfunction
Mortality rate | 24 weeks
  the patients' death rate related to treatment and transplantation with in 24 weeks after treatment
Acute rejection | 24 weeks
  the frequency of acute rejection
Progression to albuminuria | 24 weeks
  the frequency of macroalbuminuria
Progression to macroalbuminuria | 24 weeks
  the frequency of macroalbuminuria
Fasting plasma glucose | 24 weeks
  Change from baseline in fasting plasma glucose
Glycated hemoglobin (HbA1c) | 24 weeks
  Change from baseline in HbA1c
Adverse events | 24 weeks
  Record adverse events that related to treatment and transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Ni, Dr., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Shan Mou, Dr., Study Director — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Yaomin Hu, Dr., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Ming Zhang, Dr., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Department of nephrology, endocrinology and kidney transplantation , Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882